CLINICAL TRIAL: NCT01556009
Title: A Phase II Randomized, Open Label Trial Comparing the Effects of Intermittent Vismodegib Versus PDT on the Maintenance of Benefit Following 7 Months of Continuous Vismodegib Treatment in Patients With Multiple Basal Cell Carcinomas
Brief Title: Trial Comparing the Effects of Intermittent Vismodegib vs. PDT in Patients With Multiple Basal Cell Carcinomas
Acronym: Vismodegib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-077; ML28244 (Other Grant/Funding Number: Genentech)
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Basal Cell Nevus Syndrome; Gorlin's Syndrome
Keywords: Basal Cell Carcinoma; Photodynamic Therapy
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Carcinoma, Basal Cell | interventions — HhAntag691; Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug (Vismodegib) (Active Comparator): Vismodegib taken orally 150 mg per day for 7 continuous months then randomized for 3 month intervals to 28 months.
  Interventions: Drug: Vismodegib
- Aminolevulinic acid %20 topical solution (Active Comparator): Aminolevulinic acid HCL 20% topical solution applied every three months from month 10, 13, 16, 19, 22. Applied and incubated for three hours.
  Interventions: Drug: Aminolevulinic acid %20 topical solution

INTERVENTIONS:
Drug: Vismodegib — 150 mg per day for 7 continuous months then randomized for 3 month intervals to 28 months.
  Other Names: Erivedge; GDC-0449
  Arms: Drug (Vismodegib)
Drug: Aminolevulinic acid %20 topical solution — 20% topical solution applied every three months from month 10, 13, 16, 19, 22. Applied and incubated for three hours.
  Other Names: Levulan
  Arms: Aminolevulinic acid %20 topical solution

SUMMARY:
The purpose of this study is to evaluate and compare the safety and efficacy of intermittent vismodegib and of Photodynamic Therapy (PDT).

DETAILED DESCRIPTION:
This is a Phase II, 28 month, randomized, two arm multicenter clinical study design. During the initial 7 months of the study, all 24 subjects will receive vismodegib, 150mg/day. They then will be randomized in a 1:1 ratio to receive intermittent vismodegib, 150 mg/day, during months 10-13, 16-19, and 22-25 or to receive treatment with PDT at month 10 and at three month intervals thereafter. The safety and efficacy of intermittent vismodegib and of PDT will be assessed at the time of the subjects' visits to the Study Center and at the time of telephone contacts. A Data Safety Monitoring Board (DSMB) will review results for an interim analysis when 12 subjects have completed 28 months. The DSMB review will focus on adverse events and efficacy results. Subjects will be monitored for the presence of surrogate endpoint biomarkers (SEBs) at each Study visit.

ELIGIBILITY:
Inclusion Criteria:

The subject:

* has had diagnosed at least 10 SEB (of diameter 3 mm diameter or greater on the nose or periorbital skin, 5 mm or greater elsewhere on the face, or 9 mm or greater on non-facial areas excluding the skin below the knees) during the two years before study entry.
* meet diagnostic criteria for basal cell nevus syndrome
* is willing to abstain from application of non-study topical medications to the skin for the duration of the study. For example, topical preparations containing corticosteroids (other than Triamcinolone applied no more than 6x/month).
* is willing to forego treatment of BCCs unless the BCCs are documented by Study Investigators, preferably on two separate visits, except when the PSCP believes that delay in treatment potentially might compromise the health of the subject.
* has normal laboratory tests as defined by the following: Normal hematopoietic capacity, Normal hepatic function: AST and ALT greater than or equal to 2x the upper limit of normal (ULN) Total bilirubin within normal range 0.20 mg/dl to 1.50 mg/dl or within 3x ULN for patients with Gilbert's disease Normal renal function: normal serum creatinine or measured creatinine clearance less than 50 mL/minute. Fasting cholesterol greater than or equal to 220 untreated
* be willing to not donate blood or semen for three months following discontinuation of Study medications.
* is willing to avoid pregnancy in his partner as defined by the following: Male subject is willing to use a latex condom during the study and for 3 months after the last dose during sexual contact with a female of childbearing potential, even if he has had a successful vasectomy. His partner must also use a form of birth control

Exclusion Criteria:

The subject:

* has used topical or systemic therapies that might interfere with the evaluation of the study medication during the study. Specifically these include the use of: (i) glucocorticoids (other than Triamcinolone on no more than 36 days during the six months prior to study entry) to more than 5% of the skin (ii) retinoids systemically or topically to more than 5% of the skin during the six months prior to study entry; (iii) alpha-hydroxy acids to more than 5% of the skin during the six months prior to study entry (iv) 5-fluorouracil or imiquimod systemically or topically to the skin above the knees during the six months prior to study entry. (v) treatment with systemic chemotherapy within one year prior to starting study medication.
* has a history of hypersensitivity to any of the ingredients in the study medication formulations.
* is unable to return for follow-up visits and tests.
* has uncontrolled systemic disease, including known HIV positive patients.
* has history of congestive heart failure.
* has uncontrolled hypocalcemia, hypomagnesemia, or hypokalemia
* has clinically important history of liver disease, including viral or hepatitis, current alcohol abuse, or cirrhosis.
* has any condition or situation which in the Investigator's opinion may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study.
* has a history of invasive cancer within the past five years excluding non-melanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of the breast, or CLL Stage 0.
* has current, recent (within 4 weeks of Day 1), or planned participation in an experimental drug study while enrolled in this study.
* is a female who is pregnant, plans to ever to become pregnant, capable of becoming pregnant or is breast feeding.
* is a male who is unwilling or unable to comply with pregnancy prevention measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Epstein, MD, Principal Investigator — Children's Hospital Research Institute
Locations (3):
- United States (3):
  - Children's Hospital Oakland Research Institiute, Oakland, California
  - Children's Hospital Research Center Oakland, Oakland, California
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has left the institution and sincere efforts were made to contact the PI, but were unsuccessful. No data are available to report.
Period: Overall Study
Arm/Group | Drug (Vismodegib) | Aminolevulinic Acid %20 Topical Solution
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and sincere efforts were made to contact the PI, but were unsuccessful. No data are available to report.
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug (Vismodegib) | Aminolevulinic Acid %20 Topical Solution | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence to Baseline SEB Burden Following 7 Months of Continuous Vismodegib Treatment.
Description: Primary:
  i. To compare the efficacy of (i) intermittent vismodegib vs. (ii) the efficacy of photodynamic therapy (PDT) in preventing the return of the burden of surgically eligible BCCs (SEBs) to baseline level following 7 months of continuous vismodegib therapy.
  ii. To compare the cumulative diameter (burden) of SEBs in patients treated intermittently with vismodegib vs. with photodynamic therapy (PDT).
Time Frame: A Data Safety Monitoring Board (DSMB) will review results for an interim analysis when 12 subjects have completed 28 months.
Population: as for baseline characteristics
Arm/Group | Drug (Vismodegib) | Aminolevulinic Acid %20 Topical Solution
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Cumulative Diameter (Burden) of SEBs in Patients Treated Intermittently With Vismodegib vs PDT During Months 8-28 Maintenance Period.
Description: i. To assess the safety of intermittent vismodegib in patients with multiple BCCs (BCNS and non-BCNS) during months 8-28.
  ii. To assess resistance of SEBs to treatments in patients with multiple BCCs (BCNS and non-BCNS) treated intermittently during months 8-28.
  iii. To assess the degree of reduction of SEBs after 7 months of continuous daily vismodegib therapy.
  iv. To conduct an exploratory evaluation in non-BCNS patients with multiple BCCs (high burden of disease) of the efficacy and tolerability of intermittent vismodegib vs PDT
Time Frame: as for outcome 1
Population: as for baseline characteristics
Arm/Group | Drug (Vismodegib) | Aminolevulinic Acid %20 Topical Solution
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The PI has left the institution and sincere efforts were made to contact the PI, but were unsuccessful. No data are available to report.
Arm/Group | Drug (Vismodegib) | Aminolevulinic Acid %20 Topical Solution
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes